CLINICAL TRIAL: NCT04259398
Title: The Influence of Type of Anesthesia on Mortality and Cancer Recurrence After Colon Cancer Surgery: Multi-center Prospective Randomized Controlled Study
Brief Title: Anesthesia and Cancer Study: Colon Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Korean Society of Anesthesiologists (Unknown); Seoul National University Bundang Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Seoul St. Mary's Hospital (Other); Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor (full), Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ane-Can colon (1912-133-109)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Cancer of Colon; Anesthesia
Keywords: anesthesia; propofol; cancer; inhalational anesthetics
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA (Experimental): propofol infusion targeting bispectral index 40-60
  Interventions: Drug: Propofol
- inhalation (Sevoflurane) (Active Comparator): sevoflurane targeting bispectral index 40-60
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — propofol 1-2 mg/kg bolus injection for induction of anesthesia propofol continuous infusion for maintenance of anesthesia
  Arms: TIVA
Drug: Sevoflurane — sevoflurane is administered for induction and maintenance of anesthesia
  Arms: inhalation (Sevoflurane)

SUMMARY:
This study investigates the influence of type of anesthesia on survival and recurrence rate in patients receiving colon cancer surgery. The participants will be allocated to either the TIVA group and the inhalation group.

DETAILED DESCRIPTION:
The effect of anesthesia on cancer recurrence and survival is controversial. According to some retrospective studies and preclinical studies, total intravenous anesthesia (TIVA) is suggested to be more favorable than inhalation anesthesia regarding cancer recurrence and survival after surgery. However, there is no randomized controlled study to determine this difference in colon cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* adults undergoing surgery to remove colon cancer

Exclusion Criteria:

* pregnancy
* colon cancer with invasion to perineum
* palliative surgery
* history of diagnosis or surgery for other cancer
* emergent surgery
* ASA PS classification 4 and 5
* refusion to participate in the study
* allergy to anesthetics

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 797 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2028-05-03 (Estimated); Study Completion 2028-05-03 (Estimated)

PRIMARY OUTCOMES:
five year survival | five years survival
  survival rate regardless of recurrence

SECONDARY OUTCOMES:
five year recurrence free survival | five years after surgery
  survival rate without recurrence
1 year recurrence free survival | 1 year after surgery
  survival rate without recurrence
3 year recurrence free survival | 3 years after surgery
  survival rate without recurrence
1 year survival | 1 year after surgery
  survival regardless of recurrence
3 year survival | 3 years after surgery
  survival regardless of recurrence

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No